CLINICAL TRIAL: NCT04128072
Title: MOGAT: Open-Label, Phase II, Multi-Centre, Study of Anti-CCR4 Monoclonal Antibody (Mogamulizumab) and Total Skin Electron Beam Therapy (TSEB) in Patients With Stage IB-IIB Cutaneous T-Cell Lymphoma
Brief Title: Anti-CCR4 Monoclonal Antibody (Mogamulizumab) and Total Skin Electron Beam Therapy (TSEB) in Patients With Stage IB-IIB Cutaneous T-Cell Lymphoma
Acronym: MOGAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1820-CLTF
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Stage IB-IIB Cutaneous T-Cell Lymphoma
Keywords: Cutaneous T-Cell Lymphoma; Mogamulizumab; Total Skin Electron Beam therapy
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mogamulizumab + Total Skin Electron Beam Therapy (TSEB) (Experimental): Treatment with mogamulizumab will be continued until disease progression or the occurrence of another withdrawal criterion as specified in the protocol.
  TSEB will start 28 days after mogamulizumab cycle 2 day 1 at a dose of 12 Gy in 8 fractions over two weeks (4 fractions per week).
  Interventions: Drug: Mogamulizumab; Radiation: Total Skin Electron Beam Therapy (TSEB); Drug: Mogamulizumab (subsequent cycles post TSEB)

INTERVENTIONS:
Drug: Mogamulizumab — • Patients will receive mogamulizumab 1.0 mg/kg IV over at least 1 hour on Days 1, 8, 15 and 22 of the first 28 day treatment cycle (C1) and on Days 1 and 15 of subsequent 28 day cycle (C2).
Radiation: Total Skin Electron Beam Therapy (TSEB) — * After completion of C2, patients will be administered TSEB at a dose of 12 Gy in 8 fractions (4 fractions per week). TSEB will start 28 days (window of + 7 days) after mogamulizumab (C2 D1).
  * In case of toxicity from mogamulizumab, the maximum delay permitted for the start of TSEB is 2 weeks.
  * If recovery to at least grade 1 from toxicity exceeds the 2 weeks interval, please contact the medical monitor.
  * Mogamulizumab is stopped during TSEB administration.
Drug: Mogamulizumab (subsequent cycles post TSEB) — • Mogamulizumab will be restarted at a dose of 1.0 mg/kg IV on Days 1, 8, 15 and 22 for cycle 3. Subsequent cycles will be administered as for C2.
  Treatment with mogamulizumab will be continued until disease progression (PD) or the occurrence of another withdrawal criterion.

SUMMARY:
Cutaneous T-Cell Lymphoma (CTCL) has a chronic, relapsing course with patients undergoing multiple, consecutive therapies. Treatment aims at the clearance of skin disease, minimization of recurrence, prevention of disease progression and preservation of quality of life.

The treatment of CTCL is primarily determined by the disease extent. Prolonged complete remissions have been obtained with skin-directed therapies in early stage Mycosis fungoides (MF) (IA-IIA), whereas advanced stages CTCL (IIB-IVB) are often refractory to treatment and, thus, have an unfavorable prognosis.

Currently, there is no standard treatment option for CTCL, especially for advanced stages, and the optimal treatment sequence is still debated with a large variability in the therapeutic approach across countries. Patients with advanced-stage disease or refractory cutaneous CTCL should be treated with systemic therapies and, whenever possible, should be offered to participate in clinical trials. Currently, there is a urgent call for new treatments in CTCL with higher response rate and prolonged time to progression;

In this study, we propose a very innovative treatment schedule in which mogamulizumab is used before Total Skin Electron Beam therapy (TSEB) for systemic disease control and as a maintenance treatment after skin-directed therapy. We hypothesize that our regimen will show a more manageable toxicity profile than a combination treatment and allow for a long-term mogamulizumab administration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MF stage IB, IIA or IIB at registration, and MF stage should have never met criteria for stage IIIA or higher.
* Subjects who have failed (refractory or relapsed) at least one prior course of systemic therapy.
* All clinically significant toxic effects of prior cancer therapy to grade ≤ 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE, v.5.0), excluding the specifications required in the criteria 'Adequate haematological and organ function' below
* Males and female subjects ≥ 18 years
* WHO performance status 0-1
* Adequate haematological and organ function:
* absolute neutrophil count (ANC) ≥ 1.0 × 109/L
* platelets ≥ 75 × 109/L (≥ 75,000/mm3)
* bilirubin ≤ 1.5 × upper limit of normal (ULN) except for subjects with Gilbert's syndrome;
* aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN
* serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance > 50 mL/min using the Cockcroft-Gault formula
* Subjects previously treated with anti-CD4 antibody or alemtuzumab are eligible provided a washout period ≥ 3 months and CD4+ cell counts ≥ 200/mm3
* Clinically normal cardiac function based on 12-lead ECG and above the institutional lower limit of normal for left ventricular ejection fraction assessed either by multi-gated acquisition scan or cardiac ultrasound
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 3 days prior to the first dose of study treatment
* WOCBP must agree to use effective contraception, defined as oral contraceptives, double barrier method (condom plus spermicide or diaphragm plus spermicide) or practice through abstinence from sexual intercourse during the study and for 6 months after the last dose.
* Male subjects and their female partners of child bearing potential must be willing to use an appropriate method of contraception defined as oral contraceptives, double barrier method (condom plus spermicide or diaphragm plus spermicide) or practice through abstinence from sexual intercourse (periodic abstinence, e.g., calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception) during the study and for 6 months after the last dose.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* Prior treatment with mogamulizumab, or any other anti-CCR4
* Prior TSEB
* Patients who received localised radiotherapy within 2 weeks prior to registration
* Patients who received any systemic therapy for MF within 4 weeks prior to registration.

Note: In case of rapid progression, if patient has recovered from all toxicities AND last dose occurred more than 5 half lives of the drug/treatment used, patient could be allowed to start earlier after consultation with medical monitor

* History of other malignancy in the past 5 years with the exception of treated carcinoma in situ of the cervix, localized prostate cancer with PSA <0.1, in-situ melanoma, and non-melanoma skin cancer
* History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins
* Known hypersensitivity to CHO cell products or any component of the mogamulizumab formulation (see section 6.1.1)
* Significant uncontrolled intercurrent illness including, but not limited to:
* uncontrolled infection requiring antibiotics;
* clinically significant cardiac disease (class III or IV of the New York Heart Association [NYHA] classification);
* unstable angina pectoris;
* angioplasty, stenting, or myocardial infarction within 6 months;
* clinically significant cardiac arrhythmia
* Have active sign of herpes zoster
* Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
* Patients with eczema, psoriasis, lichen simplex chronicus, with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
* Rash must cover <10% of body surface area
* Disease is well controlled at baseline and requires stable use of low to mild potency topical corticosteroids for at least 4 weeks.
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 4 months.
* Immunomodulatory drugs or high-dose systemic steroids for concomitant or intercurrent conditions other than T-cell lymphoma within 7 days of registration.

However, stable dose of a low dose systemic systemic corticosteroid (≤10 mg prednisone equivalent per day) or stable dose of a low potency topical corticosteroid for at least 4 weeks prior to the registration is permitted. Subjects may receive intra-articular, intraocular, inhalation or nasal corticosteroids. Initiation of treatment with corticosteroids or increase in dose while on study is not permitted except for the treatment of adverse events.

* Patients who are planned to receive stem cell transplantation
* Has a known history of Human T-lymphotropic virus 1 (HTLV-1), or human immunodeficiency virus (HIV) (test to be performed within 21 days of registration if allowed by local legislation)
* Has known active Hepatitis B or Hepatitis C
* Note: patient will be eligible if:
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening . The HBV DNA test will be performed only for patients who have a positive total HBcAb test.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival Rate at 48 weeks | Up to 48 weeks after start of mogamulizumab for each patient
  The primary endpoint is the progression free survival rate, assessed at 48 weeks after start of mogamulizumab

SECONDARY OUTCOMES:
Occurrence of Adverse Events | 48 months after last patient in
Response rate to both mogamulizumab and TSEB | From the first patient treatment start till 48 weeks as of last patient in
  Proportion of patients achieving partial response or complete response according to EORTC-ISCL-USCLC criteria
Progression-free survival | From the first patient treatment start till 48 weeks as of last patient in
  From start of mogamulizumab to the first date of progressive disease or death from any cause
Overall survival | From the first patient treatment start till 5 years after last patient treatment
  Start of mogamulizumab till the date of death from any cause
Time to progression | From the first patient treatment start till 48 weeks as of last patient in
  From start of mogamulizumab to the date of first documentation of progressive disease or death due to progressive disease, whichever occurs first
Duration of response | From the first patient treatment start till 48 weeks as of last patient in
  Duration of response will be measured for patients achieving a partial response or complete response are first met until the first date that recurrent or progressive disease
Time to next treatment | From the first patient treatment start till 48 weeks as of last patient in
  From time from initiation of mogamulizumab until the time the initiation of any total skin-equivalent treatment (topical treatment to >50% of body surface, phototherapy, second TSEB) or systemic treatment is recorded

OTHER OUTCOMES:
Quality of life using the Skindex-29 questionnaire | 48 months after last patient in
  The Skindex-29 is a skin disease-specific questionnaire that comprehensively assesses the effects of skin diseases on patient's quality of life
Quality of life using the EORTC-QLQ-C30 questionnaire | 48 months after last patient in
  Quality of Life will be assessed by using the EORTC-QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Luis Ortiz Romero, Principal Investigator — Hospital Universitario 12 De Octubre,Madrid, Spain; Richard Cowan, Principal Investigator — The Christie NHS Foundation Trust Manchester, UK; Jan Nicolay, Principal Investigator — UniversitaetsMedizin Mannheim, Mannheim, Germany
Locations (13):
- University Hospitals Copenhagen - Rigshospitalet, Copenhagen, Denmark
- France (2):
  - CHU de Bordeaux - Groupe Hospitalier Saint-Andre - Hopital Saint-Andre, Bordeaux
  - Assistance Publique Hopitaux Paris- APHP Nord - Univ De Paris Cite - Hop. Saint Louis, Paris
- Germany (2):
  - UniversitaetsMedizin Mannheim, Mannheim
  - Muehlenkreiskliniken Johannes Wesling Klinikum Minden, Minden
- Athens University - Attikon University General Hospital, Athens, Greece
- Italy (2):
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino - Ospedale San Lazzaro, Torino
- Spain (3):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario Puerta De Hierro, Madrid
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust (UHB) -Queen Elizabeth Medical Centre, Birmingham
  - The Christie NHS Foundation Trust, Manchester